CLINICAL TRIAL: NCT06391450
Title: Study of Empagliflozin in Patients With Autosomal Dominant Polycystic Kidney Disease (EMPA-PKD)
Acronym: EMPA-PKD
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-505890-3
Record Dates: First submitted 2024-04-15; First posted 2024-04-30 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Autosomal Dominant Polycystic Kidney
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin 10 milligram (MG) (Experimental)
  Interventions: Drug: Empagliflozin 10 MG
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Oral
  Arms: Empagliflozin 10 milligram (MG)
Drug: Placebo — Oral
  Arms: Placebo

SUMMARY:
The EMPA-PKD trial is assessing the safety of empagliflozin in patients with rapid progressive ADPKD with and without concomitant tolvaptan use by monitoring kidney growth and the rate of loss of kidney function.

DETAILED DESCRIPTION:
In autosomal dominant polycystic kidney disease (ADPKD) formation of cysts in the kidneys causes destruction of functional parenchyma and loss of kidney function, which may progress to end-stage kidney disease. Tolvaptan is the only drug specifically approved for slowing down the progression of ADPKD. Sodium glucose cotransporter 2 inhibitors (SGLT2i) might provide additional benefits but there is currently no information on safety and outcome effects of SGLT2i in patients with ADPKD, as these patients were excluded in the landmark SGLT2i trials. In an investigator-initiated, double-blind, mono-center, placebo-controlled, randomized clinical trial the EMPA-PKD study is assessing the safety of empagliflozin in patients with rapid progressive ADPKD with and without concomitant tolvaptan use by monitoring kidney growth and the rate of loss of kidney function.

44 participants will be randomly allocated (1:1) to receive a daily dose of either empagliflozin (10 mg/day) or placebo for 18 months. Patients will be stratified according to concomitant tolvaptan use. The primary endpoint is progression of cystic kidney growth by monitoring MRI-based changes in total kidney volume and the secondary endpoint is exploring changes in glomerular filtration rate. Additional endpoints include adverse events and changes in copeptin levels, albuminuria and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female* patients ≥ 18 of age
2. Screening eGFR ≥ 25 and ≤ 90 mL/min/1.73 m2 if age ≥ 18 and ≤50 years or Screening eGFR ≥ 25 and ≤ 65 mL/min/1.73 m2 if age > 50 years
3. ADPKD diagnosed by unified criteria (combination of family history, ultrasound, MRI/CT, genotyping as needed)
4. Mayo Class I C, D, E
5. Patients with and without tolvaptan use will be included. Patients with tolvaptan use will be included if tolvaptan has been taken for ≥ 3 months at study entry.
6. Willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures
7. Evidence of signed written informed consent.

Exclusion criteria:

1. Kidney or any other solid organ transplant recipient
2. Currently receiving SGLT2-inhibitor
3. Concomitant treatment with steroids or any other immunosuppressive agent
4. Hypersensitivity to the active principle (Empagliflozin) or any of the excipients (e.g. lactose)
5. Ketoacidosis (laboratory based) in the past 5 years
6. Type 1 diabetes mellitus
7. Ongoing urinary tract- or genital infections
8. Inability to fully understand the possible risks and benefits related to study participation
9. Inability to undergo MRI exam (e.g. implanted medical devices)
10. Women who are pregnant or breastfeeding
11. Unwilling to practice acceptable methods of birth control during study participation
12. Participation in another clinical trial (other investigational drugs or devices at the time of enrolment or within 30 days prior to enrolment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Total kidney volume (TKV) | 18 months
  Relative change from baseline TKV (percent/year) to month 18 of treatment.

SECONDARY OUTCOMES:
Estimated glomerular filtration rate (eGFR) | 18 months
  Change in the eGFR from baseline to month 18 of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Roland SCHMITT, MD, Principal Investigator — Hannover Medical School
Locations (1):
- Medizinische Hochschule Hannover, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eswarappa M, Madden E, Shlipak MG, Cui X, Mrug M, Estrella MM, Park M. Sodium-Glucose Cotransporter-2 Inhibitor Therapy and Longitudinal Changes in Kidney Function among Veterans with Autosomal Dominant Polycystic Kidney Disease. Clin J Am Soc Nephrol. 2025 May 16;20(7):940-949. doi: 10.2215/CJN.0000000725. PMID 40377984
- [Derived] Bahlmann-Kroll E, Hackl S, Kramer S, Wulfmeyer VC, Glandorf J, Kaufeld J, Koch A, Hartung D, Schmidt BMW, Schmidt-Ott K, Schmitt R. Empagliflozin in patients with autosomal dominant polycystic kidney disease (EMPA-PKD): study protocol for a randomised controlled trial. BMJ Open. 2024 Dec 15;14(12):e088317. doi: 10.1136/bmjopen-2024-088317. PMID 39675824
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039